CLINICAL TRIAL: NCT05209269
Title: Comparing Oxygen Saturation Stability and Work of Breathing Between Normal Term Infants and Premature Infants Prior to Discharge
Brief Title: Work of Breathing in Term Infants
Status: Completed | Type: Observational
Sponsor: Christiana Care Health Services (Other)
Responsible Party: Sponsor
Other Study IDs: DDD605112
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2023-09-11 (Actual); Status verified 2023-09

CONDITIONS: Work of Breathing; Term Infant

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Work of breathing observation — We will place soft elastic bands around the infant's chest and abdomen to assess their work of breathing.

SUMMARY:
This is a prospective observational cohort study conducted in the mother-baby unit at ChristianaCare. The study is designed to assess work of breathing indices and oxygen saturation stability at discharge in full-term infants. Data obtained will be used to perform a comparative analysis on work of breathing data for premature infants obtained from our previous study. We hypothesize full term (≥37 weeks gestation) infants have decreased work of breathing indices (i.e., phase angle) compared to premature infants (born 26-37 weeks gestation) at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Infants born ≥37 weeks gestation
* Admitted to the Mother-Baby Unit
* Within 24 hours of expected discharge

Exclusion Criteria:

* Infants born between < 37week gestation admitted to the Mother-Baby Unit at CCHS
* Infants with skeletal, neuromuscular, or abdominal surgical disorders that affect the accuracy of work of breathing measurements will also be excluded.

Ages: 1 Day to 1 Week | Sex: All
Age Groups: Child
Study Population: Infants born ≥37 weeks gestation admitted to the Mother-Baby Unit
Sampling Method: Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2022-04-22 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Work of breathing indices | 25 minutes
  A phase angel of 0 represents perfect synchrony between the chest and abdominal compartments. Higher phase angles represent greater degrees of asynchronous breathing. A phase angle of ≥ 40 represents asynchrony and increased work of breathing. A phase angle of 180 represents complete asynchrony.

SECONDARY OUTCOMES:
Oxygen saturations | 25 minutes
  Oxygen saturations will be measured by the high-resolution pulse oximeter.

CONTACTS AND LOCATIONS:
Overall Officials: Kelley Z Kovatis, MD, Principal Investigator — Christiana Care Health Services
Locations (1):
- Christiana Care Health Services, Inc., Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: No
De-identified data will be shared with our statistical colleagues. Published data will be in aggregate form.